CLINICAL TRIAL: NCT02339506
Title: Stress and the Nervous System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Gail Kurr Adler, Associate Professor, Brigham and Women's Hospital
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: 2014P002423
Record Dates: First submitted 2015-01-06; First posted 2015-01-15 (Estimated); Results first posted 2017-11-30 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Autonomic Nervous System; Baroreflex; Stress, Physiological
Keywords: stress; ACTH; cosyntropin; baroreflex sensitivity; cardiovagal
MeSH Terms: interventions — Cosyntropin; Adrenocorticotropic Hormone; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cosyntropin (Active Comparator): Subjects will receive cosyntropin infusion at 70 mcg/hr for two sessions of 2.5 hours each on day 2 of a three day admission to our research center.
  Interventions: Drug: Cosyntropin
- Normal saline (Placebo) (Placebo Comparator): Subjects will receive normal saline infusion for two sessions of 2.5 hours each on day 2 of a three day admission to our research center.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cosyntropin — Subjects will receive cosyntropin at 70 mcg/hr for two sessions of 2.5 hours each on day 2 of a three day admission to our research center.
  Other Names: ACTH
  Arms: Cosyntropin
Drug: Placebo — Subjects will receive placebo (normal saline infusion) for two sessions of 2.5 hours each on day 2 of a three day admission to our research center.
  Other Names: Normal Saline
  Arms: Normal saline (Placebo)

SUMMARY:
Models of stress such as hypoglycemia have identified that stress results the next day in decreased baroreflex sensitivity. This project will test the hypothesis that these delayed changes in autonomic nervous system function are secondary to a rise in ACTH. The investigators will infuse cosyntropin versus placebo in a double-blind, crossover study in healthy adults and measure the delayed effects on the autonomic system as measured by cardiovagal baroreflex sensitivity.

DETAILED DESCRIPTION:
Stress has complex effects on the body's physiology. Models of stress such as hypoglycemia have identified that stress activates the hypothalamic-pituitary-adrenal (HPA) axis and sympathoadrenal system acutely. Additionally, there are delayed effects of prior exposure to hypoglycemia. The day after being exposed to a hypoglycemic stimulus there are: 1) decreases in the catecholamine release to a new hypoglycemic stress; 2) decreases in the muscle sympathetic nerve activity (MSNA) response to either a new hypoglycemic challenge or transient hypotension; 3) decreases in cardiac vagal baroreflex sensitivity (BRS); and 4) increases in sensitivity to thermal pain and altered temporal summation (decreased tolerance to a repeated minimally painful stimulus). This project will test the hypothesis that these delayed changes in autonomic nervous system function are secondary to a rise in ACTH that occurs in response to stress.

Primary Aim. Infusion of ACTH (cosyntropin) will lead the next day to decreased cardiovagal baroreflex sensitivity in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

Subjects must be currently healthy, BMI 18-32 kg/m2, and not be on any medications.

This study will recruit men and women. Due to concerns about estrogen's effects on hormone levels and possible contributions of menstrual symptoms on pain sensing thresholds, we will schedule the inpatient studies to avoid the early follicular phase in normally cycling women.

Subjects must have normal laboratory values for:

1. Complete blood count
2. Serum creatinine, sodium, potassium, glucose, liver enzymes
3. Urinalysis
4. Urine pregnancy test (if female)
5. Normal ECG

Exclusion Criteria:

We will exclude individuals with:

* Systolic blood pressure > 140 or < 90 mm Hg
* Diastolic blood pressure > 90 mm Hg
* Creatinine clearance ≤ 60 mL/min, as calculated by MDRD formula
* Known DM, CHF, CAD, PVD, CVA, MI, asthma
* Known or history of Cushing's disease or adrenal insufficiency
* Known neurologic disease
* Known psychiatric disease
* Steroid use (oral or inhaled, local or systemic injections, within the past 6 months)
* Significant concomitant medical illnesses
* Current excessive alcohol (>10oz ethanol/week)
* Current use of recreational drugs
* Current smokers
* Current pregnancy
* Chronic use of non-steroidal anti-inflammatory or narcotic medications
* Evidence of ischemia or heart block on screening electrocardiogram (greater than type I-second degree heart block, left bundle branch block, or ST-T wave changes in 2 or more contiguous leads)
* Subjects taking any prescription medications (other than oral birth control pills) or herbal medications will be excluded.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2020-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gail Adler, MD, PhD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Zaheer S, Meyer K, Easly R, Bayomy O, Leung J, Koefoed AW, Heydarpour M, Freeman R, Adler GK. Effect of adrenocorticotropic hormone infusion on circulating sclerostin levels. Endocr Connect. 2021 Dec 14;10(12):1607-1614. doi: 10.1530/EC-21-0263. PMID 34788228
- [Derived] van der Boom T, Jia C, Lefrandt JD, Connelly MA, Links TP, Tietge UJF, Dullaart RPF. HDL Cholesterol Efflux Capacity is Impaired in Severe Short-Term Hypothyroidism Despite Increased HDL Cholesterol. J Clin Endocrinol Metab. 2020 Sep 1;105(9):e3355-62. doi: 10.1210/clinem/dgaa411. PMID 32761088
- [Derived] Leung JH, Bayomy OF, Bonyhay I, Celli J, White J, Freeman R, Adler GK. ACTH Infusion Impairs Baroreflex Sensitivity-Implications for Cardiovascular Hypoglycemia-Associated Autonomic Failure. J Clin Endocrinol Metab. 2020 Jul 1;105(7):2345-53. doi: 10.1210/clinem/dgaa221. PMID 32353115

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo (Period 1)/Washout (Period 2)/Cosyntropin (Period 3): Period 1: Subjects will receive a placebo infusion for two sessions of 2.5 hours each on day 2 of their first three day admission to our research center.
  Period 2: Washout for one month Period 3: Subjects will receive cosyntropin infusion at 70 mcg/hr for two sessions of 2.5 hours each on day 2 of their second three day admission to our research center.
- Cosyntropin (Period 1)/Washout (Period 2)/ Placebo (Period 3): Period 1: Subjects will receive a cosyntropin infusion at 70 mcg/hr for two sessions of 2.5 hours each on day 2 of their first three day admission to our research center.
  Period 2: Washout for one month Period 3: Subjects will receive a placebo infusion for two sessions of 2.5 hours each on day 2 of their second three day admission to our research center.
Period: Period 1 (Placebo or Cosyntropin)
Arm/Group | Placebo (Period 1)/Washout (Period 2)/Cosyntropin (Period 3) | Cosyntropin (Period 1)/Washout (Period 2)/ Placebo (Period 3)
Started | 12 | 11
Completed | 12 | 10
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Period: Washout (Period 2)
Arm/Group | Placebo (Period 1)/Washout (Period 2)/Cosyntropin (Period 3) | Cosyntropin (Period 1)/Washout (Period 2)/ Placebo (Period 3)
Started | 12 | 10
Completed | 10 | 10
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0
Period: Period 3 (Placebo or Cosyntropin)
Arm/Group | Placebo (Period 1)/Washout (Period 2)/Cosyntropin (Period 3) | Cosyntropin (Period 1)/Washout (Period 2)/ Placebo (Period 3)
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Arm/Group | Healthy Control
Number analyzed (Participants) | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 23
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 22
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 14
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Cardiovagal Baroreflex Sensitivity (Modified Oxford Technique)
Description: Cardiovagal baroreflex sensitivity will be measured with the Modified Oxford Technique before, during, and after drug infusions, to evaluate the effects of cosyntropin infusions.
Time Frame: Baseline, 4-hours after infusion, 24-hours after infusion
Measure: Mean (Standard Deviation); unit: ms/mmHg
Arm/Group | Cosyntropin | Normal Saline (Placebo)
Number analyzed (Participants) | 20 | 20
ms/mmHg
  Baseline | 17.75 (5.47) | 16.90 (8.63)
  4-hours after infusion | 14.42 (5.89) | 17.27 (6.79)
  24-hours after infusion | 14.76 (5.83) | 18.90 (8.40)

2. Other Pre Specified Outcome: Pain (Quantitative Sensory Testing Using a Thermal Pain Testing Device)
Description: Alterations in pain sensing will be evaluated pre and post with quantitative sensory testing using a thermal pain testing device, to evaluate the delayed effect of cosyntropin infusions.
Time Frame: 1 day after ACTH
Reporting Status: Not Posted

3. Other Pre Specified Outcome: Hippocampal Memory (Paired Associative Learning Task)
Description: Hippocampal memory will be evaluated pre and post with a paired associative learning task. Face Name Associative Memory Exam (FNAME) composite score on a scale from 0-36, with 36 being the best possible score.
Time Frame: 1 day after ACTH
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cosyntropin | Normal Saline (Placebo)
Number analyzed (Participants) | 20 | 20
score on a scale
  Baseline | 27.8 (3.7) | 29.3 (2.8)
  1 day after infusion | 25.6 (4.1) | 25.9 (4.1)

ADVERSE EVENTS:
Arm/Group | Placebo | Cosyntropin
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/21
Other Adverse Events (participants affected / at risk) | 2/22 | 0/21
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=22) | Cosyntropin (N=21)
vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) — Subject vomited during study, likely due to GI illness.
Subject had less blood drawn (General disorders) | 1 (1) | 0 (0) — Subject with normal Hct at screen (37.8), had low Hct on admission (30.8 and 31.9). Due to general wellness the study proceeded; blood draws were reduced to primary endpoints/safety and only about 40cc of blood were drawn (reduced from about 165 cc).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No